CLINICAL TRIAL: NCT00626639
Title: A Phase 1/2 Study to Evaluate Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of Weekly Doses of Palifermin (rHuKGF) for the Reduction of Oral Mucositis in Subjects With Locally Advanced Head and Neck Cancer (HNC) Receiving Postoperative Radiotherapy With Concurrent Chemotherapy
Brief Title: A Study of Palifermin for the Reduction of Oral Mucositis in Patients With Locally Advanced Head and Neck Cancer Receiving Postoperative Radiotherapy and Concurrent Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20040124; NCT00963378 (obsolete NCT alias)
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-05

CONDITIONS: Mucositis; Head and Neck Cancer
Keywords: palifermin; Clinical Trial; Oncology; Head & Neck
MeSH Terms: conditions — Mucositis; Head and Neck Neoplasms; Neoplasms | interventions — Fibroblast Growth Factor 7; Radiotherapy; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Three days before the start of radiotherapy (Day -3), participants received a single intravenous (IV) bolus injection of matching placebo. During radiotherapy (beginning on Day 1), participants received a weekly single IV bolus injection of matching placebo after the last radiation fraction of that week (usually on Fridays) until grade ≥3 oral mucositis occurred, or for a maximum 8 doses (completion of radiotherapy). Participants also received cisplatin 100 mg/m^2 on days 1, 22 and 43.
  Interventions: Drug: Placebo; Radiation: Radiotherapy; Drug: Cisplatin
- Palifermin (Experimental): Three days before the start of radiotherapy (Day -3), participants received a single intravenous (IV) bolus injection of palifermin at 120 μg/kg. During radiotherapy (beginning on Day 1), participants received a weekly single IV bolus injection of palifermin at 120 μg/kg after the last radiation fraction of that week (usually on Fridays) until grade ≥3 oral mucositis occurred, or for a maximum 8 doses (completion of radiotherapy). Participants also received cisplatin 100 mg/m^2 on days 1, 22 and 43.
  Interventions: Drug: palifermin; Radiation: Radiotherapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Placebo — Administered by intravenous (IV) bolus injection
  Arms: Placebo
Drug: palifermin — Administered by intravenous (IV) bolus injection
  Arms: Palifermin
Radiation: Radiotherapy — Once daily irradiation of 20 centigray (cGy)/day x 33 fractions for a total target dose of 6600 cGy (conventional radiation therapy using standard fractionation [one fraction per day])
Drug: Cisplatin — 100 mg/m^2 intravenously (IV) on days 1, 22 and 43.

SUMMARY:
Oral Mucositis associated with adjuvant radiation and concurrent chemotherapy in postoperative Head and Neck setting

DETAILED DESCRIPTION:
This study consisted of 2 phases. The acute oral mucositis (OM) evaluation phase includes the time from randomization to the time of severe OM (WHO Grade 3 or 4) resolution (up to Week 12 or up to Week 15 for participants whose severe OM is not resolved at Week 12). In the acute OM evaluation phase, participants were randomized to receive either a single IV bolus dose of palifermin or placebo at 120 μg/kg, 3 days before the start of radiotherapy, plus 7 once-weekly palifermin or placebo doses at the same dose level during a 7-week radio/chemotherapy course. In the long-term follow up phase, participants are followed until death, withdrawal of consent, or loss to follow-up. The long-term follow up phase is still ongoing.

ELIGIBILITY:
Inclusion Criteria:

* History of newly diagnosed histologically confirmed squamous cell carcinoma (American Joint Committee on Cancer [AJCC] Stage II, III, IVA, or IVB) involving either the oral cavity, oropharynx, nasopharynx, hypopharynx, or larynx, post surgical resection (R0, R1)
* Scheduled to receive adjuvant concurrent chemoradiation treatment within 12 weeks of surgery
* High-risk subject defined by presence of at least one of the following: R1 resection margins; T3 or T4 tumor stage; 3 or more positive lymph node metastases; <3 lymph node metastases with extracapsular extension of the disease
* Radiation treatment field to receive planned dose of at least 50Gy to areas of the oral cavity/oropharynx mucosa that can be visualized

Exclusion Criteria:

* Tumors of the lips, paranasal sinuses, salivary glands, or of unknown primary tumors
* Metastatic disease (M1) / Stage IV C
* Presence or history of any other primary malignancy
* History of pancreatitis
* Prior radiotherapy to the site of disease
* Prior chemotherapy
* Other investigational procedures
* Thirty days or less since receiving an investigational product or device in another clinical trial. Current enrollment in another clinical trial is not permitted unless the sole purpose of the trial is for long-term follow-up/survival data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-07; Primary Completion 2007-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After recruitment of 5 participants, the study was closed to further enrollment due to administrative changes at the study center (ie, departure of principal investigator) and slow enrollment.
Period: Overall Study
Arm/Group | Placebo | Palifermin
Started | 2 | 3
Completed | 0 (Participants who received all 8 doses of investigational product.) | 1 (Participants who received all 8 doses of investigational product.)
Not Completed | 2 | 2
Not completed — Occurrence of grade 3 oral mucositis | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Palifermin | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Median (Full Range); unit: years] | 53.0 [38 to 68] | 52.0 [44 to 65] | 52.0 [38 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event is an undesirable medical occurrence (sign, symptom, or diagnosis) or worsening of a pre-existing medical condition occurring after start of study drug up to the end of acute oral mucositis (OM) evaluation phase, whether or not considered to be study drug related. If severe OM was not resolved by Week 12, AEs were documented until resolution of severe OM or Week 15, whichever occurred first. A serious AE is any event that is fatal, life threatening, requires or prolongs hospitalization, is a persistent or significant disability/incapacity or is a congenital anomaly/birth defect. The intensity of AEs was graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v3 based on the following: Grade 1 = Mild AE, Grade 2 = Moderate AE, Grade 3 = Severe AE, Grade 4 = Life-threatening or disabling AE, Grade 5 = Death related to AE. A Protocol-specific Limiting Toxicity (PSLT) is any non-hematologic Grade 3 or 4 AE considered related to study drug.
Time Frame: Up to Week 12 (or Week 15 for participants with severe OM was not resolved by Week 12)
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 2 | 3
participants
  Any adverse event | 2 | 3
  Serious adverse event | 0 | 2
  Severe AE (Grade 3, 4 or 5) | 0 | 2
  Treatment related adverse event | 0 | 1
  Treatment related serious AE | 0 | 1
  Treatment related severe AE (Grade 3, 4 or 5) | 0 | 1
  Study Discontinuation Due to AE | 0 | 0
  Protocol Specific Limiting Toxicity (PSLT) | 0 | 0
  Deaths | 0 | 1

2. Primary Outcome: Ratio of Ki67-positive Cells Before and After Palifermin Treatment
Description: The effect of palifermin on cell proliferation was to be assayed by staining for the cell cycle proliferation marker Ki67 in buccal mucosal biopsy samples taken prior to the first dose and either 24 or 48 hours after the first dose. Due to the small sample size, this analysis was not performed.
Time Frame: Day -3 predose and 24 or 48 hours post-dose
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Pharmacokinetics of Palifermin
Description: Due to the small sample size this analysis was not performed.
Time Frame: Day -3, predose and at 2, 5, 15, 30, 60, and 90 minutes and 2, 4, 6, 8, 10, 12, 24 and 48 hours after the first dose
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Severe Oral Mucositis (OM) (Adapted RTOG/EORTC Grade ≥3)
Description: The adapted RTOG/EORTC mucositis assessment scale as follows: Grade 0 = no change; Grade 1 = mild enanthema, mild pain; Grade 2 = patchy mucositis, moderate edema, moderate pain; Grade 3 = confluent fibrinous mucositis, massive edema, massive pain; Grade 4 = extensive ulceration, confluent necrosis, massive hemorrhage.
  Due to the small sample size this analysis was not performed.
Time Frame: Assessed daily up to Week 12 (or Week 15 if severe oral mucositis not resolved ≤ adapted RTOG/EORTC Grade 2 by Week 12).
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Patient-Reported Mouth and Throat Soreness Score
Description: The average patient-reported mouth and throat soreness (MTS) score as reported on question 3 of the Oral Mucositis Questionnaire for Head and Neck Cancer [OMQ-HN]): "How much mouth and throat soreness did you experience in the past 24 hours?" Participants answered on a scale from 0 (no soreness) to 4 (extreme soreness).
  Due to the small sample size this analysis was not performed.
Time Frame: Assessed daily up to Week 12 (or Week 15 if severe oral mucositis not resolved ≤ adapted RTOG/EORTC Grade 2 by Week 12).
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Disease Progression by Week 12
Description: Disease progression was determined by clinical examination and histopathologic examination by the Investigator.
Time Frame: Up to Week 12
Population: Tumor response data was missing for one participant.
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 2 | 2
participants | 1 | 0

7. Secondary Outcome: Overall Survival
Description: Deaths during long-term follow up of subject participating in the acute phase of the study receiving placebo or Palifermin.
Time Frame: During long-term follow-up phase, until December 2015
Population: Subjects who received placebo duringthe acute phase of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Subjects who received placebo during the acute phase of the study.
- Palifermin: Subjects who received Palifermin during the acute phase of the study.
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 2 | 3
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: Up to 15 weeks from first dose of IP
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo | Palifermin
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2) | Palifermin (N=3)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Red blood cell count increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Gum neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2) | Palifermin (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Oral pain (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Bacteriuria (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Pharmacokinetic, pharmacodynamic, safety and efficacy endpoints were not evaluable due to the limited number of subjects enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits sponsor a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Sponsor may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, investigator agrees not to publish any results before the first multi-center publication.